CLINICAL TRIAL: NCT04599699
Title: A Phase I Integrated Boost to the Dominant Intraprostatic Nodule Based on Ga-68 Prostate-Specific Membrane Antigen (PSMA) PET/MR Study of Stereotactic Body Radiation Therapy in Patients With Localized Prostate Cancer
Brief Title: Integrated Boost to the Dominant Intraprostatic Nodule Based on Ga-68 PSMA PET/MR Study of SBRT With Prostate Cancer
Acronym: SBRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Clinical Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Changhai Hospi
Record Dates: First submitted 2020-10-10; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Treatment
Keywords: SBRT; prostate cancer; Ga-68 PSMA PET/MR
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Androgen Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Simultaneously integrated boost or sequential integrated boost
  * Simultaneously integrated boost Prostate tumor: starting dose 8.7 Gy per fraction in 5 fractions (total 43.5 Gy) Prostate gland: fixed prophylactic tumoricidal dose 7.25 Gy per fraction in 5 fractions. Total 36.25 Gy.
  * Sequential integrated boost Prostate tumor: starting dose 7.25 Gy per fraction in 6 fractions (total 43.5 Gy) Prostate gland: fixed prophylactic tumoricidal dose 7.25 Gy per fraction in 5 fractions. Total 36.25 Gy.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Very Low, Low, favorable, or Good Prognostic Intermediate prostate cancer:SBRT; Unfavorable, or Poor Prognostic Intermediate prostate cancer: SBRT accompanied 4 months ADT;High or Very High prostate cancer: SBRT accompanied 2 years ADT.
  Other Names: androgen deprivation therapy (ADT)

SUMMARY:
The aim of this study is to test the safety and efficacy of integrated boost to the dominant intraprostatic nodule based on Ga-68 Prostate-Specific Membrane Antigen (PSMA) PET/MR in Stereotactic Body Radiation Therapy (SBRT) in localized prostate carcinoma in patients for whom the standard treatment is the irradiation of the entire prostate gland with or without seminal vesicles accompanied or not by hormonal therapy.

DETAILED DESCRIPTION:
Radiotherapy is considered standard of care treatment for prostate cancer. In light of the accumulating clinical evidence favoring the use of hypo fractionation, SBRT regimen might constitute a much more convenient non-invasive and highly efficient outpatient therapy. Although the proposed extreme hypofractionated radiotherapy approach was expected to provide excellent local control of the primary prostate cancer, a proportion of patients with intermediate- or high-risk disease may have recurrences with local recurrence or distant metastasis in the future, requiring strategies to minimize systemic disease. Ga-68 PSMA PET/MR has high accuracy in the diagnosis and staging of prostate cancer. In this protocol, pretreatment Ga-68 PSMA PET/MR and CT scanning were performed in all patients as well as the imaging fusion before delineating the target. This study would explore the simultaneously integrated boost or equential integrated boost to the dominant intraprostatic nodule based on Ga-68 PSMA PET/MR in SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* tumor clinical stage cT1-3N0M0 according to AJCC TNM 2017
* Without any treatment of prostate cancer including radiotherapy, ADT, chemotherapy, focal treatment, etc.
* With the examination of Ga-68 PSMA PET/MR
* International Prostate Symptom Score(IPSS）<15 (alpha blockers allowed), without severe urethral obstruction symptoms
* ECOG performance status 0-2
* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures

Exclusion Criteria:

* Prior pelvic RT
* A tumor located at less than 3 mm from the urethra or rectum when measured at the MRI
* Tumor clinical stage cT4, with metastases including bone, lymph nodes or organ metastasis
* Histologically confirmed neuroendocrine tumor or small cell carcinoma of the prostate
* Severe or active co-morbidity likely to impact on the advisability of SBRT like severe liver or kidney dysfunction, etc.
* Patients with other malignancies, or acute or other severe infections, with ulcerative colitis, inflammatory bowel disease, etc.
* Patients who have participated in other clinical trials for less than three months
* Patients have acute prostatitis or chronic prostatitis with urinary symptoms
* Urine routine indicates obvious urinary system infection and no significant improvement after anti-infective treatment, or conversion to recurrent urinary system infection
* Unsuitable to participate in this clinical trial judged by the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The Probability of Acute genitourinary (GU) , gastrointestinal (GI) toxicity and erectile dysfunction | 90 days after the first fraction of radiotherapy treatment
  Acute genitourinary (GU) , gastrointestinal (GI) toxicity and erectile dysfunction (ED) (grade 2 or more) according to the NCI CTCAE v4.0.

SECONDARY OUTCOMES:
The Probability of Chronic genitourinary (GU) , gastrointestinal (GI) toxicity and erectile dysfunction (ED) | > 90 days and up to 3 years from the start of protocol treatment
  Chronic genitourinary (GU) , gastrointestinal (GI) toxicity and erectile dysfunction (ED) (grade 2 or more) according to the NCI CTCAE v4.0.
1-year Biochemical Progression-free Survival (bPFS) | Assessment at 1-year
  Biochemical Progression-free Survival (bPFS)
1-year Local Progression-Free-Survival(LPFS) | Assessment at 1-year
  Local Progression-Free-Survival(LPFS)
1-year Distant Metastasis Free Survival(DMFS) | Assessment at 1-year
  Distant Metastasis Free Survival(DMFS)
1-year Overall Survival (OS) | Assessment at 1-year
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao X, Zhu X, Cheng C, Jiang L, Ye Y, Cao Y, Li Y, Zuo C, Zhang H. Protocol of the integrated boost to the dominant intraprostatic nodule in stereotactic body radiation therapy for localized prostate cancer. Future Oncol. 2022 Dec 12. doi: 10.2217/fon-2022-0590. Online ahead of print. PMID 36507781